CLINICAL TRIAL: NCT02219022
Title: Progressive Resistance Exercise in Rheumatoid Arthritis Patients: a Randomized Controlled Trial
Brief Title: Progressive Resistance Exercise in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Felipe Martinelli Lourenzi, PT, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP/UNIFESP 1826/10
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Progressive resistance exercise; Pain; Functional capacity; Quality of life; Muscle strength
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Patient remain with their usual clinical treatment.
  Interventions: Other: Control group
- Experimental group (Experimental): Patients in experimental group participated in a 12-week progressive resistance training using a maximum repetition exercise in which patients performed 1 Maximum Repetition with the maximum bearable weight. Once the 1 Maximum Repetitionwas determined, training was divided into the following regimen: 2 series of 8 repetitions, the first with 50% and the second with 70% of 1 Maximum Repetition.
  The exercises were knee extension and flexion and hip abduction and adduction, elbow extension and flexion, wrist extension and flexion and shoulder abduction and adduction and spine extension and flexion all performed in machines. The 1 Maximum Repetition load was reevaluated every 6 weeks.
  Patient remain with their usual clinical treatment.
  Interventions: Other: Control group; Other: Experimental group

INTERVENTIONS:
Other: Control group
  Other Names: Clinical tretament
Other: Experimental group
  Arms: Experimental group

SUMMARY:
A randomized controlled trial with rheumatoid arthritis patients will be realized. Patients will be randomized into two groups. Experimental group will do a 12 weeks training of progressive resistance exercise for global muscles and remain with the clinical treatment and the control only remain with the clinical treatment. Patients will be evaluated at baseline, after 6, 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to American College of Rheumatology 2010
* Both genders
* Age between 18 and 65 years
* Functional class I, II and III
* Stable medication within the three months preceding the study
* Haven't done any kind of regular exercise (two or more times per Week) for at least three months before study start
* Have agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Participating in another type of study
* Have difficulty understanding the evaluation tools with fibromyalgia
* Joint deformities that make impossible do the exercises
* Other musculoskeletal diseases
* Other diseases that contraindicate exercises.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in pain - Visual analogue scale | baseline, 6, 12 and 24 weeks

SECONDARY OUTCOMES:
Change in function capacity - Health Assessment questionaire | Baseline, after 6, 12 and 24 weeks
Change in quality of life - Short form 36 | baseline, after 6, 12 and 24 weeks
Change in strength - 1 maximum repetition | baseline, after 6, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil